CLINICAL TRIAL: NCT00547599
Title: Does Presence of Distress Due to Erectile Dysfunction Affect the Effect of Tadalafil on Sexual Life and Life Satisfaction?
Brief Title: Determine If the Stress That Comes With Not Developing an Erection Affects Tadalafil Effects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7989; H6D-SO-LVFR
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): 20 mg tadalafil tablet
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 20 mg tadalafil tablet by mouth as needed, no more than once a day for 8 weeks.
  Other Names: LY450190; Cialis; IC351

SUMMARY:
To determine if patients who are distressed over having problems getting or maintaining an erection react differently to the medication than those who are not stressed over the issue.

ELIGIBILITY:
Inclusion Criteria:

* 3 months history of erectile dysfunction (ED)
* Anticipate a monogamous relationship with a female sexual partner
* Be able to make minimum required sexual intercourse attempts
* Abstain from using any other ED treatment

Exclusion Criteria:

* Nitrate use
* Participated in previous tadalafil study or have a current tadalafil prescription
* Heart attack within the last 90 days
* Kidney problems
* Certain heart problems

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2003-04; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Change In Spontaneity Domain of PAIRS scale scores | 8 weeks

SECONDARY OUTCOMES:
Change in the Time Concerns, Sexual Self-Confidence & Sexual Miscommunication, domains of PAIRS scale scores | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uppsala, Sweden

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com